CLINICAL TRIAL: NCT03863769
Title: The Influence of Chiropractic Distraction Spinal Manipulation on Posture and Performance in Patients With Lumbar Spinal Stenosis.
Brief Title: Chiropractic Distraction Spinal Manipulation- Lumbar Stenosis Study
Acronym: Stenosis
Status: Completed | Type: Observational
Sponsor: Parker University (Other)
Collaborators: University of Houston (Other); Whittier College (Unknown); Private Practice (Unknown); Miami University (Other)
Responsible Party: Sponsor
Other Study IDs: Parker19_02
Record Dates: First submitted 2019-02-14; First posted 2019-03-05 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Chiropractic manipulation; postural sway; distraction manipulation; performance-based mobility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Lumbar Spinal Stenosis: Questionnaire, chiropractic treatment, and posture and performance testing.
  Interventions: Other: Lumbar Spinal Stenosis

INTERVENTIONS:
Other: Lumbar Spinal Stenosis — Posture and Performance testing: ABC-6 Scale, low back pain NRS, buttock or leg pain NRS, five times sit-to-stand, timed up-and-go, PGIC, eyes open force plate assessment (30 seconds), and eyes closed force plate assessment (30 seconds).

SUMMARY:
To assess the effect of chiropractic distraction manipulation on postural sway and simple measures of performance in patients with the clinical diagnosis of lumbar spinal stenosis.

DETAILED DESCRIPTION:
This study aims to assess the effect of chiropractic distraction manipulation in reducing postural sway and improving performance-based mobility and disability in patients with the clinical diagnosis of lumbar spinal stenosis. This study will identify if distraction spinal manipulation will reduce postural sway center of pressure (COP) movements as determined by a force plate, if distraction spinal manipulation will improve simple measures of performance-based mobility and if distraction spinal manipulation will improve perception of balance confidence and will reduce self-rated stenosis associated disability.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 48 years old
* Patient has leg or buttock pain while walking
* Patient feels relief of symptoms with bending (flexing) forward
* Patient feels relief when using a shopping cart of bicycle
* Patient has motor or sensory disturbance while walking
* Patient has normal and symmetrical foot pulses
* Patient has lower extremity weakness
* Patient has low back pain
* Duration of symptoms and signs for more than 1 month
* Able to stand and walk without assistive devices for at least 20 minutes
* Able to give written informed consent and complete interviews and questionnaires in English

Exclusion Criteria:

* Complicated spinal pain due to fracture, tumor, infection, or severe spondyloarthropathy
* Has other severe co-morbidities, including progressive neurological deficit
* Other serious pathologies of the locomotor system
* No correspondence availability through email
* Inability to read/ comprehend English
* Compensation or seeking compensation from a third-party liability or workers' compensation
* Previous spinal manipulation within the past month

Min Age: 48 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population studied will be existing and/or new patients at the Cox Certified Doctor's private practice.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Balance tracking | Each participant will be tested for one minute
  The primary outcome is static balance as assessed by center of pressure (COP) using a portable force plate (Balance Tracking Systems, BTrackS™).

SECONDARY OUTCOMES:
Questionnaire: Pain sclae | 5 Minutes
  Pain severity of the lower back and buttock using a numerical rating scale (0-10)
Questionnaire: Disability | 5 Minutes
  Stenosis specific disability using the Zurich Claudication Questionnaire; symptom and function. Zurich Claudication Questionnaire has a 7-item symptom severity subscale with scores from 1 to 5 and a 5-item physical function subscale with scores from 1 to 4. The total score range is 12 to 55 points, with higher scores indicating higher levels of self-reported disability.
Questionnaire: Balance | 5 Minutes
  Balance Specific Confidence (ABC-6)
Questionnaire: Change | 5 Minutes
  Patient Global Impression of Change, this 1-item question has a 7-point rating scale with 1 being no change and 7 being considerable improvement.
Sit to Stand | 5 Minutes
  physical performance as assessed by the 5 Times Sit to Stand and Timed Up and Go tests.

CONTACTS AND LOCATIONS:
Overall Officials: Katie Pohlman, DC, MS, PhD, Principal Investigator — Parker University
Locations (1):
- Parker University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Information about this study and individual data will be made available per request and approval from all investigator members.
Supporting Information: Study Protocol, ICF, CSR